CLINICAL TRIAL: NCT02113072
Title: Recurrent Wheezing in Infants: Risk Factors and Prevention With Probiotics, a Randomized Clinical Trial, Double-blind, Placebo Controlled.
Brief Title: Recurrent Wheezing in Infants: Risk Factors and Prevention With Probiotics.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Geórgia Véras de Araújo, Postgraduate in Allergy and Clinical Immunology., Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAraujo
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Tract Diseases; Wheezing
Keywords: wheezing, immune system, cytokines, probiotics, infants.
MeSH Terms: conditions — Respiratory Tract Diseases; Respiratory Sounds | interventions — Beclomethasone; Probiotics; Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics & Beclomethasone (Experimental): It will be supplied in lyophilized form, in each sachet containing 1 g of the probiotic, to be used in addition to milk, juice or yoghurt in the first morning meal once daily for 60 days.
  Beclomethasone HFA 50mcg spray - 100 mcg/day as initial treatment for primary and wheezing in this age group, at doses considered minimal, for 4 months.
  Interventions: Drug: Beclomethasone; Drug: Probiotics
- Beclomethasone & Placebo (Active Comparator): The placebo will be supplied in the same way with the same organoleptic characteristics of formula with probiotics. It will be supplied in lyophilized form in each sachet containing 1 g of placebo, to be used in addition to milk, juice or yoghurt in the first morning meal once daily for 60 days.
  Interventions: Drug: Beclomethasone; Drug: Placebo

INTERVENTIONS:
Drug: Beclomethasone — The wheezing infants will be using the inhaled corticosteroid beclomethasone 50mcg - 02 jets per day (100mcg/dia).
  Other Names: Clenil
Drug: Probiotics — Lyophilized form, each sachet containing 1 g of the probiotic, to be used in addition to milk, juice or yoghurt in the first morning meal once daily for 60 days.
  Other Names: Lactobacillus; Bifidobacterium; Leveduras; Acetobacter
  Arms: Probiotics & Beclomethasone
Drug: Placebo — The placebo will be supplied in the same way with the same organoleptic characteristics of formula with probiotics, 1 g sachet for 60 days, in the juice, milk or yoghurt.
  Other Names: Maltodextrose
  Arms: Beclomethasone & Placebo

SUMMARY:
The purpose of this study is to evaluate whether Probiotics promote reduction of recurrent wheezing in infants, stimulating the immune system to Th1 response.

DETAILED DESCRIPTION:
OBJECTIVES

GENERAL

* Assess whether probiotic supplementation reduces the frequency of recurrent wheezing in infants .

SPECIFIC

* Identifying the presence of environmental and genetic factors to recurrent wheezing in infants, which may serve as major confounders of the effect of probiotics in the sample studied risk factors .
* Check the effect of probiotics as the recurrence of wheezing in infants.
* Evaluate the effects of probiotics on the immune response of the infant wheezing , through the measurement of IL - 10 , IL - 12 and Interferon-gama before and after intervention with the use of probiotics .

DESIGN RESEARCH

Study Design

* Inferential, the type longitudinal, randomized trial, double-blind, parallel, placebo-controlled study.

Intervention to be held:

* Patients attended at the Infant Hospital of the Federal University of Pernambuco will undergo clinical investigation and completion of baseline examinations is eligible to participate in the study after informed consent from parents or guardians. Infants with recurrent wheezing, six months to two years of age, will be divided into two groups - one receiving the formula with probiotics (treatment group) and the other formula with similar organoleptic characteristics, placebo (control group).

Flowchart of randomization

* Patients assessed for eligibility verification will be randomized and follow the CONSORT flowchart second Guide - 2011.

IMPLEMENTATION OF RESEARCH

Local and survey period

* Hospital das Clinicals, Federal University of Pernambuco - UFPE, Brazil. Period April 2014 to Abril 2015.

Population Research

* Method of Selection of Sample
* Sample selection of recurring wheezing infants attended at Infant Hospital das Clinicas UFPE, to be considered eligible for admission to the study and meet the criteria for inclusion and exclusion. The wheezing infants selected as eligible for the study remained with wheezing even using inhaled corticosteroids.

Type of Randomization and Allocation Mechanism

* A simple randomization of patients will be by draw of numbers 1 - 60.

Randomization was performed by a third person who used a randomization program on the computer.

The sequence of random numbers, recruitment and allocation of patients to the intervention by the principal investigator of the study will be conducted.

Sample Size

* The sample size calculation was based on two studies on probiotics and asthma, whereas a level of less than 5% , a power study of 80% and an acceptable error of up to 20%, 60 patients significance can be sufficient to analyze the number of desired effect evaluation of wheezing in infants and reject or accept the null hypothesis.

Operationalization Steps

* The infants were considered eligible for the study, will have the free and informed consent to participate in the study signed by their parents and or guardians.

These patients initially attended, shall undergo a medical examination protocol with questions and answers QE - EISL (technical interview with the parents or guardians) and achievement of immediate skin test sensitivity to major aeroallergens and food allergens (mites, cat and dog epithelium, molds, feathers, cockroaches, egg yolk, egg white and cow's milk proteins) through the skin prick test and chest radiography.

Patients before starting probiotics or placebos, will the dosage of the cytokines IL-10, IL-12 and INF-gamma, IgE and eosinophils.

The wheezing infants will be using the inhaled corticosteroid beclomethasone 50mcg - 02 jets per day (100mcg - dia), found this medication for free, brand name and specifications: Clenil HFA 50mcg spray 200 doses as initial and fundamental treatment for wheezing this age group, at doses considered minimal.

The formula with probiotics containing 10 CFU (Colony Forming Unit)/g consortium of probiotic strains of lactobacilli, lactococcus, streptococcus, yeasts and acetobacter type in appropriate concentrations per gram. It will be supplied in lyophilized form, in each sachet containing 1 g of the probiotic, to be used in addition to milk, juice or yoghurt in the first morning meal once daily. The placebo will be supplied in the same way with the same organoleptic characteristics of formula with probiotics.

During this period, the infant wheezing present crisis, parents or guardians will note the day of wheezing attacks and treatment used in a standardized form with open answers, which will be provided, and will contact you by telephone, with the researcher. Parents or guardians will receive a daily record of control, to assess the occurrence of wheezing attacks.

After eight weeks of using probiotics, infants will undergo new measurement of cytokines IL - 10 , IL - 12 and Interferon - gama, with the objective to evaluate the immune response of probiotics in both groups.

Before and at the end of each period, the patient will undergo physical examination and parents or guardians to an interview, to assess the occurrence of wheezing attacks.

These data will be analyzed to assess whether supplementation with probiotics reduces the frequency of wheezing in infants.

Masking and Allocation Mechanism

A third member of the study will assign a number to probiotics and placebo recipients in accordance with the numbers of randomization, without the knowledge of the investigator and the patient. Containers should be equal and contain substances of the same organoleptic characteristics. The containers will be provided in numerical order, as service and previous randomization.

Instruments Measurement and Assessments

QE- EISL: written questionnaire (International Study of Wheezing in Infants) - see Appendix 01, which is an instrument consisting of 45 questions on demographic characteristics, wheezing and its potential risk factors. Originally developed in Spanish, was translated into Portuguese (Brazilian) and validated. This protocol will be used with closed questions with answers, using the technical interview, conducted by the researcher, the parents or guardians.

Statement of Informed Consent Form (ICF) - see apêncice 02 - after approval thereof in having their children participating in the study.

Control plug - clinical - see Appendix 03: will be used by parents or guardians to describe the date, " wheezing " and perceived treatment need, while using the probiotic or placebo (08 weeks) and 08 weeks more.

Prick Test: standardized extracts dihiclorada histamine (10mg/ml) and 0.9% saline (FDA - Immunotech , Rio de Janeiro , Brazil) will be used. The extracts will be dripped on the volar surface of the forearm and then performed one puncture with sterile lancet. As a positive control we histamine and negative saline control. The diameter of each reaction will be evaluated after 15 minutes and the result expressed as positive if wheal ≥ 3mm negative control.

Eosinophil count and total serum IgE Dosage: will be held in peripheral blood collection vessel with qualified professional lab, in the amount of 7.0 ml. The reference values are appropriate for age and standardization of laboratory.

Chest radiography: held at the radiology department of the Hospital das Clinicals - UFPE.

Dose of IL - 10 , IL - 12 and Interferon-gama: will be held in peripheral blood collection vessel with qualified professional lab in the amount of 5.0 ml. This blood will be taken to the Laboratory Ageu Magalhães, which will be submitted to centrifugation and performed by the supernatant of peripheral blood mononuclear cells (PBMC), the count of cytokines in serum. Then the cultivation of these cells for 48 hours and subsequent counting of cytokine IL - 10 , IL - 12 and Interferon - gama is performed.

The peripheral blood mononuclear cells at a concentration of 1 x 106 cells/mL are collected from the patients of the treatment group and the placebo group and are incubated with phytohemaglutinin (PHA ; 10μg/ml) for 48 hours. Production of IL - 10, IL - 12 and Interferon - gama in culture supernatant will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits. The detection limit for these cytokines will be 5ρg/ml .

STATISTICAL ANALYSIS

Statistical Methods for Data Analysis

* For statistical analysis Initially , a probability distribution (percent analysis) is performed. Subsequently, the techniques of normal distribution and homogeneity of variances by means of ShapiroWillks and bartlett, respectively, tests will be applied to characterize the use of the parametric Student's t tests or Manny Whitney for independent samples. For categorical variables the chi- square test for association with Yates correction will be used. Data are expressed as mean and standard deviation ( parametric test ) or median and standard error ( nonparametric test ) with a significance level of p < 0.05 . 21 for Windows 2011 - to generate the analyzes , the statistical package SPSS will be used.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged six months to two years incomplete.
* Infants who have recurrent wheezing in the past 3 months.
* Infants under use of proper technique of inhaled corticosteroids: beclomethasone HFA spray - 50 mg - 2 times daily (100 mg / day) with spacer and face mask.

Exclusion Criteria:

* Patients who present congenital airway malformations, cystic fibrosis, chronic diseases in other systems, perinatal respiratory problems, allergy to the protein in cow's milk, intrathoracic tumors, Tuberculosis and Pulmonary Congenital immunodeficiencies, children who were premature: <37 weeks gestational age.
* Use of other products containing probiotics in its composition with previous exposure or even study period.
* Infant in use of anti-leukotrienes.
* Use recent antibiotic.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Recurrent wheezing and cytokine assay. | After 2 months of using probiotic, will be assessed the recurrence of wheezing and cytokine assay.
  After eight weeks of using probiotics, infants will undergo new measurement of cytokines IL-10, IL-12 and INF-γ, with the objective to evaluate the immune response of probiotics in both groups.
  Before and at the end of each period, the patient will undergo physical examination and parents or guardians to an interview, to assess the occurrence of wheezing attacks.
  These data will be analyzed to assess whether supplementation with probiotics reduces the frequency of wheezing in infants.

CONTACTS AND LOCATIONS:
Overall Officials: Geórgia V. Araújo, Doctor, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Rose MA, Stieglitz F, Koksal A, Schubert R, Schulze J, Zielen S. Efficacy of probiotic Lactobacillus GG on allergic sensitization and asthma in infants at risk. Clin Exp Allergy. 2010 Sep;40(9):1398-405. doi: 10.1111/j.1365-2222.2010.03560.x. Epub 2010 Jun 28. PMID 20604800
- [Background] Kopp MV, Hennemuth I, Heinzmann A, Urbanek R. Randomized, double-blind, placebo-controlled trial of probiotics for primary prevention: no clinical effects of Lactobacillus GG supplementation. Pediatrics. 2008 Apr;121(4):e850-6. doi: 10.1542/peds.2007-1492. Epub 2008 Mar 10. PMID 18332075
- [Background] Ozdemir O, Erol AY. Preventative and therapeutic probiotic use in allergic skin conditions: experimental and clinical findings. Biomed Res Int. 2013;2013:932391. doi: 10.1155/2013/932391. Epub 2013 Sep 1. PMID 24078929 (Retraction: PMID 24971365 Biomed Res Int. 2014;2014:965213)
- [Background] Ozdemir O. Any role for probiotics in the therapy or prevention of autoimmune diseases? Up-to-date review. J Complement Integr Med. 2013 Aug 6;10:/j/jcim.2013.10.issue-1/jcim-2012-0054/jcim-2012-0054.xml. doi: 10.1515/jcim-2012-0054. PMID 23921494
- [Background] Isolauri E, Rautava S, Salminen S. Probiotics in the development and treatment of allergic disease. Gastroenterol Clin North Am. 2012 Dec;41(4):747-62. doi: 10.1016/j.gtc.2012.08.007. PMID 23101685
- [Background] Roessler A, Forssten SD, Glei M, Ouwehand AC, Jahreis G. The effect of probiotics on faecal microbiota and genotoxic activity of faecal water in patients with atopic dermatitis: a randomized, placebo-controlled study. Clin Nutr. 2012 Feb;31(1):22-9. doi: 10.1016/j.clnu.2011.08.012. Epub 2011 Oct 2. PMID 21963389
- [Background] Azad MB, Coneys JG, Kozyrskyj AL, Field CJ, Ramsey CD, Becker AB, Friesen C, Abou-Setta AM, Zarychanski R. Probiotic supplementation during pregnancy or infancy for the prevention of asthma and wheeze: systematic review and meta-analysis. BMJ. 2013 Dec 4;347:f6471. doi: 10.1136/bmj.f6471. PMID 24304677
- [Background] Abrahamsson TR, Jakobsson T, Bjorksten B, Oldaeus G, Jenmalm MC. No effect of probiotics on respiratory allergies: a seven-year follow-up of a randomized controlled trial in infancy. Pediatr Allergy Immunol. 2013 Sep;24(6):556-61. doi: 10.1111/pai.12104. Epub 2013 Jul 31. PMID 23902407
- [Background] West CE, Hammarstrom ML, Hernell O. Probiotics in primary prevention of allergic disease--follow-up at 8-9 years of age. Allergy. 2013 Aug;68(8):1015-20. doi: 10.1111/all.12191. Epub 2013 Jul 30. PMID 23895631
- [Background] Ismail IH, Licciardi PV, Tang ML. Probiotic effects in allergic disease. J Paediatr Child Health. 2013 Sep;49(9):709-15. doi: 10.1111/jpc.12175. Epub 2013 Apr 11. PMID 23574636